CLINICAL TRIAL: NCT01395407
Title: Phase I Trial of Stereotactic Radiosurgery Following Surgical Resection of Intra-axial Brain Metastases
Brief Title: Phase I Trial of Stereotactic Radiosurgery Following Surgical Resection of Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ian Crocker, MD, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00049695; RADONC1962-11 (Other: Other)
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Brain Metastasis; Neoplasm
Keywords: Brain; Neoplasm; Neoplasm Metastasis; Radiosurgery
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A (Experimental): Cohort A: resection cavity volume up to 4.2 cc (corresponds to 0 - 2 cm diameter).
  Dose level Cohort A (Gy)
  1. 21
  2. 23
  3. 25
  Interventions: Radiation: Radiosurgery dose escalation
- Cohort B (Experimental): Cohort B: resection cavity volume > 4.2 cc and ≤ 14.1 cc (2 - 3 cm diameter).
  Dose level Cohort B (Gy)
  1. 18
  2. 20
  3. 22
  Interventions: Radiation: Radiosurgery dose escalation
- Cohort C (Experimental): Cohort C: resection cavity volume > 14.1 cc and ≤ 35 cc (3 - 4 cm diameter).
  Dose level Cohort C (Gy)
  1. 15
  2. 17
  3. 19
  Interventions: Radiation: Radiosurgery dose escalation

INTERVENTIONS:
Radiation: Radiosurgery dose escalation — Cohort A: resection cavity volume up to 4.2 cc (corresponds to 0 - 2 cm diameter).
  Cohort B: resection cavity volume > 4.2 cc and ≤ 14.1 cc (2 - 3 cm diameter) Cohort C: resection cavity volume > 14.1 cc and ≤ 35 cc (3 - 4 cm diameter)
  Dose level Cohort A (Gy) Cohort B (Gy) Cohort C (Gy)
  1. 21 18 15
  2. 23 20 17
  3. 25 22 19

SUMMARY:
Brain metastases are the most common adult intracranial tumor, occurring in approximately 10% to 30% of adult cancer patients, and represent an important cause of morbidity and mortality in this population. The standard of care for solitary brain metastasis is surgery followed by whole brain radiation therapy (WBRT). Without WBRT, there are unacceptably high levels of local failure that occur. Local recurrence rates ranged from approximately 45% at 1 year to 60% at 2 years after resection alone. However, aside from improvements in intra-cranial control, it is well documented that WBRT is associated with serious long term side effects, including significant decline in short term recall by as early as 4 months after treatment.

Many centers are now offering patients stereotactic radiosurgery (SRS) to the cavity after resection alone to improve local control while avoiding the negative effects of WBRT. There have been several retrospective studies on the use of SRS to the resection cavity alone, from which the 1 year actuarial local control rates range from 35% - 82%. The high rate of in-field local failure suggests that the current dosing regimen used may not be high enough for adequate local control. Currently, the highest local control rates are approximately 80%, but there may be room for improvement with increased dose without significantly increasing the risk of side effects.

The investigators propose a trial for patients after surgical resection of solitary brain metastases. The purpose of this trial will be to determine the maximum tolerated dose for single fraction SRS to the resection cavity. There will be three groups based on the resection cavity size. Dose escalation enrollment will be done sequentially within each cohort. You will know which cohort and which specific dose level you are randomized to. After treatment, which will take one day, regardless of cohort, you will be followed closely for treatment outcome and possible side effects. You will be asked to complete three quick surveys at each follow-up appointment regarding quality of life and memory in addition to standard of care surveillance brain MRI and physical exam.

DETAILED DESCRIPTION:
Brain metastases are the most common adult intracranial tumor, occurring in approximately 10% to 30% of adult cancer patients, and represent an important cause of morbidity and mortality in this population. The risk of developing brain metastases differs with different primary tumor histologies, with lung cancer accounting for approximately one half of all brain metastases. The prognosis of patients with brain metastases is poor. The median survival time of untreated patients is approximately 1 month. With treatment, the overall median survival time after diagnosis is approximately 4 months. The Radiation Therapy Oncology Group (RTOG) recursive partitioning analysis (RPA) describes three prognostic classes, defined by age, Karnofsky Performance Score (KPS), and disease status. The most widely used treatment for patients with multiple brain metastases is whole brain radiation therapy (WBRT). The appropriate use of WBRT can provide rapid attenuation of many neurological symptoms, improve quality of life, extend median survival, and be especially beneficial in patients whose brain metastases are surgically inaccessible or when other medical considerations preclude surgery. The use of adjuvant WBRT after resection or stereotactic radiosurgery (SRS) has been proven to be effective in terms of improving local control of brain metastases, and thus, the likelihood of neurological death is decreased.

The standard of care for solitary brain metastasis is surgery followed by WBRT. In a study by Patchell et al. for solitary brain metastases status post resection, the addition of whole brain radiation significantly reduced local recurrence from approximately 45% to 10% after resection. Although it does not prolong survival or functional independence, this treatment regimen was shown to result in significantly improved loco-regional control. A more recent study from the European Organization for Research and Treatment of Cancer (EORTC) randomized patients who underwent gross total resection (GTR) of up to 3 brain metastases to adjuvant WBRT versus observation. Adjuvant WBRT resulted in significantly reduced intracranial failure and neurologic death, however again both overall survival and functionally independent survival were not different. Among the major findings of both of these studies are the unacceptably high levels of local failure that occur after GTR alone. Local recurrence rates ranged from approximately 45% at 1 year to 60% at 2 years after resection.

However, aside from improvements in intra-cranial control, it is well documented that WBRT is associated with serious long term side effects, including significant neurocognitive decline. A randomized study conducted by Chang et al of SRS versus SRS + WBRT for 1 - 3 brain metastases found that addition of WBRT was associated with significantly worse memory recall as early as 4 months. A conclusion of this study was that a regimen of close surveillance and SRS as necessary is preferred over SRS + WBRT because the neurocognitive effects of WBRT may actually be worse than that caused by intracranial disease recurrence.

Many centers are now offering patients SRS to the cavity after resection alone to improve local control while avoiding the negative effects of WBRT. There have been several retrospective studies on the use of SRS to the resection cavity alone, from which the 1 year actuarial local control rates range from 35% - 82%. The radiation necrosis rates from these same studies range from 2% - 6%. In currently unpublished data from Emory University reviewing 63 patients with 65 cavities treated between 01/2007 and 08/2010, the 1 year actuarial local control rate was 78%. Of the 10 local failures, 70% were in-field only, 10% were marginal only, and 20% were both. The high rate of in-field failure suggests that the current dosing regimen used may be insufficient for optimal local control. The current SRS dose constraints used are derived from the phase I trial RTOG 90-05. This study determined the maximum tolerated dose for SRS in previously irradiated patients with unresected brain metastases based on lesion size. The maximum doses currently used may be artificially low for resected patients for several reasons. First, the patient population studied had been previously irradiated which most likely lowered the maximum tolerated dose versus a non-irradiated population. Secondly, the typical planning target volume (PTV) of the resection bed is the cavity with a 1 - 2mm margin. This means that the vast majority of the irradiated PTV is not brain parenchyma, but actually cerebrospinal fluid (CSF), which should result in a lower radiation necrosis rate for the same dose/volume. Currently, the highest local control rates are approximately 80%, but there may be room for improvement with increased dose without significantly increasing the risk of radiation necrosis.

The investigators propose a prospective phase I trial for patients status post surgical resection of solitary brain metastases. The purpose of this trial will be to determine the maximum tolerated dose for single fraction SRS to the resection cavity. The investigators believe that the current SRS dosing constraints may be too low, and that a larger therapeutic window exists for this patient population. Results from this trial may form the basis of future trials directly comparing WBRT with SRS to the cavity alone following resection of solitary brain metastases. This phase III study would answer the question about as to whether local irradiation is adequate treatment for patients following surgery for metastatic brain disease. Also it is anticipated that QOL measures would be built into the study in an attempt to confirm the data reported by Chang that WBRT is associated with a significant decline in QOL at even early endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic proven diagnosis of solid tumor malignancy
* Age ≥ 18
* RPA class I or class II
* Mini Mental Status Exam (MMSE) ≥ 18 prior to study entry
* Karnofsky Performance Status ≥ 70%
* Single brain metastasis status post surgical resection with ≤ 1 cc of residual enhancing tumor
* Up to 2 additional intact brain metastases to be treated with stereotactic radiosurgery (SRS) alone
* Resection cavity volume on planning scan of ≤ 35 cc
* First presentation of brain metastases
* Post-operative MRI within 72 hours of surgical resection

Exclusion Criteria:

* Previous brain radiotherapy (SRS or WBRT)
* RPA class III
* Resection cavity volume > 35 cc
* Radiosensitive or non-solid (eg. small cell lung carcinomas, germ cell tumors, leukemias, or lymphomas) or unknown tumor histologies
* Concurrent chemotherapy (no chemotherapy starting 14 days before start of radiation to 14 days after completion of radiation)
* Evidence of leptomeningeal disease by MRI and/or CSF cytology
* Current pregnancy
* More than 8 weeks between resection and radiosurgical procedure
* No metastases to brain stem, midbrain, pons, or medulla or within 7 mm of the optic apparatus (optic nerves and chiasm)
* Inability to undergo MRI evaluation for treatment planning and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 4 months after intervention
  To assess whether treating a brain resection cavity with this stereotactic radiosurgery is safe and tolerable and to determine the maximum-tolerated radiation dose for SRS to the resection cavity alone with 4-month toxicity as assessed by the RTOG central nervous system (CNS) toxicity scale

SECONDARY OUTCOMES:
Local Control | up to 2 years after intervention
  Defined as lack of progression of disease in resection cavity as assessed by period MRI scans for up to 2 years after intervention.
Distant Control | up to 2 years after intervention
  Defined as lack of progression of disease in surrounding brain as assessed by period MRI scans for up to 2 years after intervention
Neurocognitive Outcomes | up to 2 years after intervention
  Neurocognitive assessment using the Hopkins Verbal Learning Test-Revised (HVLT-R), Mini Mental Status Exam (MMSE) and Cognitive Functioning Subscale of the Medical Outcomes Scale (MOS), administered to the patient periodically for up to 2 years after intervention.
Quality of Life | up to 2 years after intervention
  Quality of life (QOL) outcomes: using the quality of life questionnaire for the Functional Assessment of Cancer Therapy-Brain (FACT-Br) administered periodically for up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Crocker, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia

REFERENCES:
- [Background] Zimm S, Wampler GL, Stablein D, Hazra T, Young HF. Intracerebral metastases in solid-tumor patients: natural history and results of treatment. Cancer. 1981 Jul 15;48(2):384-94. doi: 10.1002/1097-0142(19810715)48:23.0.co;2-8. PMID 7237407
- [Background] Sundstrom JT, Minn H, Lertola KK, Nordman E. Prognosis of patients treated for intracranial metastases with whole-brain irradiation. Ann Med. 1998 Jun;30(3):296-9. doi: 10.3109/07853899809005858. PMID 9677016
- [Background] CHAO JH, PHILLIPS R, NICKSON JJ. Roentgen-ray therapy of cerebral metastases. Cancer. 1954 Jul;7(4):682-9. doi: 10.1002/1097-0142(195407)7:43.0.co;2-s. No abstract available. PMID 13172684
- [Background] Gaspar L, Scott C, Rotman M, Asbell S, Phillips T, Wasserman T, McKenna WG, Byhardt R. Recursive partitioning analysis (RPA) of prognostic factors in three Radiation Therapy Oncology Group (RTOG) brain metastases trials. Int J Radiat Oncol Biol Phys. 1997 Mar 1;37(4):745-51. doi: 10.1016/s0360-3016(96)00619-0. PMID 9128946
- [Background] Patchell RA, Regine WF. The rationale for adjuvant whole brain radiation therapy with radiosurgery in the treatment of single brain metastases. Technol Cancer Res Treat. 2003 Apr;2(2):111-5. doi: 10.1177/153303460300200206. PMID 12680791
- [Background] Arbit E, Wronski M, Burt M, Galicich JH. The treatment of patients with recurrent brain metastases. A retrospective analysis of 109 patients with nonsmall cell lung cancer. Cancer. 1995 Sep 1;76(5):765-73. doi: 10.1002/1097-0142(19950901)76:53.0.co;2-e. PMID 8625178
- [Background] Wen PY, Loeffler JS. Management of brain metastases. Oncology (Williston Park). 1999 Jul;13(7):941-54, 957-61; discussion 961-2, 9. PMID 10442342
- [Background] Patchell RA, Tibbs PA, Regine WF, Dempsey RJ, Mohiuddin M, Kryscio RJ, Markesbery WR, Foon KA, Young B. Postoperative radiotherapy in the treatment of single metastases to the brain: a randomized trial. JAMA. 1998 Nov 4;280(17):1485-9. doi: 10.1001/jama.280.17.1485. PMID 9809728
- [Background] Kocher M, Soffietti R, Abacioglu U, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Collette S, Collette L, Mueller RP. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. J Clin Oncol. 2011 Jan 10;29(2):134-41. doi: 10.1200/JCO.2010.30.1655. Epub 2010 Nov 1. PMID 21041710
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Mathieu D, Kondziolka D, Flickinger JC, Fortin D, Kenny B, Michaud K, Mongia S, Niranjan A, Lunsford LD. Tumor bed radiosurgery after resection of cerebral metastases. Neurosurgery. 2008 Apr;62(4):817-23; discussion 823-4. doi: 10.1227/01.neu.0000316899.55501.8b. PMID 18414136
- [Background] Soltys SG, Adler JR, Lipani JD, Jackson PS, Choi CY, Puataweepong P, White S, Gibbs IC, Chang SD. Stereotactic radiosurgery of the postoperative resection cavity for brain metastases. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):187-93. doi: 10.1016/j.ijrobp.2007.06.068. Epub 2007 Sep 19. PMID 17881139
- [Background] Roberge D, Souhami L. Tumor bed radiosurgery following resection of brain metastases: a review. Technol Cancer Res Treat. 2010 Dec;9(6):597-602. doi: 10.1177/153303461000900608. PMID 21070082